CLINICAL TRIAL: NCT01501032
Title: Inpatient Evaluation of the MD-Logic Artificial Pancreas System in Patients
Brief Title: Inpatient Evaluation of the MD-Logic Artificial Pancreas System in Patients With Type 1 Diabetes
Acronym: MD-Logic- Cont
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rmc006385ctil
Record Dates: First submitted 2011-12-14; First posted 2011-12-29 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Type 1
Keywords: Diabetes Type 1; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closed Loop Control- MD-Logic (Experimental): The MD-Logic artificial pancreas system will be used in conjunction with continuous glucose monitoring and insulin pump delivery to manage the subject's blood glucose.
  Interventions: Device: MD-logic artificial pancreas system

INTERVENTIONS:
Device: MD-logic artificial pancreas system — The MD-logic artificial pancreas system is a closed loop control system using continuous glucose monitoring (CGM)and subcutaneous insulin pump infusion to mange glucose control in individuals with type 1 diabetes

SUMMARY:
The purpose of this feasibility study is to evaluate the MDLAP (MD-Logic Artificial Pancreas system)automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes. The study will include 3 inpatient admissions (12-24 hr), which will include overnight sleep, over-bolus meal, under-bolus meal and exercise.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to evaluate the MDLAP (MD-Logic artificial pancreas system)automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes. The study will include 3 inpatient admissions (12-24 hr), which will include overnight sleep, over-bolus meal, under-bolus meal and exercise. During the the visits, meal boluses will be semi-automated, with manual meal announcement by the physician/nurse, automated bolus recommendation by the system, and automated delivery of the bolus following confirmation of the recommendation. Between-meal insulin dosing will be fully automated. Bolus confirmation by the physician/nurse will be requested by the closed loop controller only when it determines that carbohydrates may be necessary to avoid hypoglycemia following the bolus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 6 months
* Age 12 to 65 years
* Hemoglobin A1c (HbA1c) between 5.0% and 10.5%, as measured with DCA2000 or equivalent device
* For females, not currently known to be pregnant
* Demonstration of proper mental status and cognition for the study
* An understanding of and willingness to follow the protocol and sign the informed consent or assent

Exclusion Criteria:

* Diabetic ketoacidosis in the past 6 months
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* History of a seizure disorder (except hypoglycemic seizure).
* Coronary artery disease or heart failure.
* Cystic fibrosis
* Active infection
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Current use of a beta blocker medication
* Hematocrit <30%
* Use of pseudoephedrine 48 hours prior to Clinical Research Center (CRC) admission

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent of glucose values 71-180 mg/dL of combined day and night readings during the first admission visit | Day 1
Percent of subjects with blood glucose reading of 71-180 mg/dL 4 hours following the breakfast with a missed meal bolus | Day 1
  Success is defined as >=40% subjects with a blood glucose in the 71-180 mg/dL range.
Percent of subjects with blood glucose reading of 71-180 mg/dL 5 hours following the breakfast with a meal bolus 30% more than the recommended bolus amount | Day 2
  Success is defined as >=50% subjects with a blood glucose in the 71-180 mg/dL range.
Percent of subjects with a blood glucose nadir <=60 mg/dL following exercise | Day 3
  Success is defined as less than 25% of subjects with a blood glucose nadir <=60 mg/dL.
Overall frequency of hypoglycemia | day 3
  Success defined as no subjects with severe hypoglycemia with a low blood glucose resulting in seizure, unconsciousness or the inability to treat oneself.
Overall frequency of hyperglycemia | Day 3
  Success defined as no subjects with diabetic ketoacidosis (DKA).
Percent of subjects with a peak blood glucose >400 mg/dL following the breakfast with a meal bolus 30% more than the recommended bolus amount | day 2
  Success is defined as less than 5% of subjects have a peak blood glucose >400 mg/dL

SECONDARY OUTCOMES:
Percent of blood glucose values 71-180 mg/dL during the day (9:00AM-11:00PM) of the first admission visit | Day 1
Percent of blood glucose values 70-180 mg/dL during the night (11:00PM-8:00AM) of the first admission visit | Day 1
Percent of blood glucose values >400 mg/dL during the first admission visit | Day 1
  Individual success is defined as no blood glucose values >400 mg/dL.
Percent of blood glucose values <=60 mg/dL during the first admission visit | Day 1
  No more than 33% of visits with blood glucose <=60 mg/dL
Percent of subjects with a peak blood glucose >400 mg/dL following the breakfast with a missed meal bolus | Day 1
  Success is defined as less than 5% of subjects have a peak blood glucose >400 mg/dL
Percent of subjects with a nadir blood glucose <=60 mg/dL following the breakfast with a missed meal bolus | Day 1
  Success is defined as less than 15% of subjects have a nadir blood glucose <=60 mg/dL
Percent of subjects with a nadir blood glucose <=60 mg/dL following the breakfast with a meal bolus 30% more than the recommended bolus amount | Day 2
  Success is defined as less than 25% of subjects have a nadir blood glucose <=60 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider children's Medical center, Petah Tikva, Israel